CLINICAL TRIAL: NCT04815564
Title: Use of Clear Aligners for the Treatment of Dental Malocclusion in Individuals With Osteogenesis Imperfecta
Brief Title: Clear Aligners for the Treatment of Dental Malocclusion in OI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of California, Los Angeles (Other); McGill University (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Brendan Lee, Professor and Chairman, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H48518
Record Dates: First submitted 2021-03-09; First posted 2021-03-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blinded to the participant information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Subjects with a PAR score between 15 and 50 and fulfilling the other eligibility criteria will be offered participation in the trial.
  Interventions: Device: Invisalign
- Natural History (No Intervention): Subjects with a PAR score outside of 15-50 will be offered the opportunity to remain on study for the Natural History arm.

INTERVENTIONS:
Device: Invisalign — Invisalign clear aligner system
  Arms: Intervention

SUMMARY:
Misalignment of teeth and jaws (also called malocclusion) is a common life altering problem facing many individuals with Osteogenesis Imperfecta (OI). The presence of Dentinogenesis Imperfecta in teeth of OI individuals makes the use of conventional orthodontics in the form of braces very challenging. Clear aligners are newer form of orthodontic treatment and is less invasive than braces. Therefore, the aim of our study is to evaluate the efficiency and safety of using Invisalign clear aligners for orthodontic treatment in individuals with Osteogenesis Imperfecta. We seek individual with Osteogenesis Imperfecta, with mild to moderate malocclusion and no prior history of orthodontic treatment. This study will be held at three sites - McGill University, University of California Los Angeles and National Institute of Dental and Craniofacial research. This study will for the first time, help define guidelines for safe and efficient orthodontic treatment using clear aligners in individuals with Osteogenesis Imperfecta. If successful, this approach can rapidly be implemented into clinical practice, as the Invisalign system is readily available to orthodontists.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is a heritable connective tissue disorder leading to frequent fractures and bone deformities. In about 90% of individuals with OI, the disease is caused by dominant mutations in one of the two genes coding for collagen type I, COL1A1 and COL1A2. The phenotype of OI ranges widely, which is captured by the Sillence classification of OI into clinical types I through IV. Individuals who have bone disease that is severe enough to lead to long-bone deformities, such as bowing of femurs and tibias, are usually diagnosed with OI type III (severe bone fragility) or IV (moderate bone fragility).

Apart from the well-known features of OI in the extracranial skeleton, OI is frequently associated with dental and craniofacial issues. These abnormalities are a source of major concern to patients. Misalignment of the jaws is a common problem in individuals with OI Type III and IV. Malocclusion associated with OI types III and IV differs markedly from the types of malocclusion commonly observed in the general population. Malocclusion in the general population is predominantly class II, however, OI types III and IV are commonly associated with class III malocclusion. The Invisalign® system (Align Technology, Santa Clara, CA) is a personalized and FDA-approved (Class II device; 510(k) number: K143630) approach to treat malocclusion. It involves incrementally moving teeth with a series of removable, custom-made clear polyurethane trays (aligners) that exert forces on teeth. The aligners are transparent ('clear aligners') and therefore are less visible than traditional braces that are made of metal. An important consideration in the treatment of patients with OI is that Invisalign does not require surface etching and cement bonding of metal braces to the tooth surface, which is difficult in the presence of dentinogenesis imperfecta. In this study, we will therefore use the Invisalign system to treat malocclusion associated with OI. This study will directly inform clinical orthodontic practice in an area of unmet clinical need and utilizes a treatment method that may be immediately implemented.

Individuals who meet the eligibility criteria will be able to enroll in the intervention arm of the study to undergo orthodontic treatment. Participants who fail to meet the eligibility criteria will be offered to participate in the study for observation purposes (natural history arm) without undergoing treatment. Participants in the intervention arm will need to visit the study site every two months for the study duration (28 months). Initial four months will involve observation period followed by two years of orthodontic treatment. Participants in the natural history arm will visit the study site every six months for a period of two years (4 visits). A complete oral exam, craniofacial evaluation, intra-oral photos, intra-oral scans, face photos, masticatory test, cone-beam CT and self-reported questionnaires will be done during the visits.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of OI.
2. Malocclusion of intermediate severity defined as a PAR score between 15 and 50.
3. Age range 12 to 40 years at the screening visit.
4. Presence of minimum number of intact teeth to proceed with orthodontic treatment.

Exclusion Criteria:

1. Prior orthodontic treatment defined as - any history of braces, palatal expansion or Invisalign treatment.
2. Candidates who meet the PAR score but need surgical intervention for correction of malocclusion
3. Presence of impacted or retained teeth.
4. Use of medication, other than bisphosphonates, known to affect bone metabolism and contraindicated on orthodontic treatment, examples are, growth hormone, corticosteroids (chronic use) and thyroid hormones.
5. Presence of other dental, oral or systemic conditions that may interfere with orthodontic treatment. Examples are severe gingivitis, active periodontal disease, cancer.
6. Pregnancy - positive during screening visit.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Peer Assessment Rating score (PAR) | Day 0, Every two months up to 28 month
  The Peer Assessment Rating (PAR) index is a valid and reliable measure of orthodontic treatment outcome and is the most widely accepted such index. A score of zero represents an ideal occlusion and in general the higher the score, the more extensive the malocclusion.

SECONDARY OUTCOMES:
Change in tooth movement | Every two months from baseline up to 24 months
  Change from baseline in anatomical tooth movement at each post-baseline time point

OTHER OUTCOMES:
QOL | Day 0 up to 28 months
  Change in Oral Health Impact Profile (OHIP-14) from the start of the observation phase to the end of the primary phase of the intervention
Masticatory efficiency | 2 month and 28 months
  Mastication expressed as number of occlusal contacts obtained from the intra-oral scans. A significant increase in the number of occlusal contacts will be interpreted as an improvement in the anatomical aspect of mastication.
Patient Satisfaction | Day 0 and up to 28months
  PSQ is a pool of 41 items assessing satisfaction with various aspects of orthodontic care. These items are paired with five-point Likert scales (1=strongly disagree, 5=strongly agree). A higher score indicates higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Lee, Principal Investigator — NIDCR/NIH; Jean-Marc Retrouvey, Principal Investigator — Baylor College of Medicine; Deborah Krakow, Principal Investigator — University of California, Los Angeles; Julia Cohen-Levy, Principal Investigator — McGill University
Locations (3):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Nidcr/Nih, Bethesda, Maryland
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No